CLINICAL TRIAL: NCT00793182
Title: A Multicenter, Double-blind, Randomized Study to Evaluate the Effects of Optiray 320 mgI/mL and Visipaque 320 mgI/mL on Renal Function in Subjects With Stable Reduced Renal Function Undergoing Contrast-enhanced Computed Tomography
Brief Title: Effects of Contrast Media on Subjects With Stable Reduced Renal Function Undergoing Contrast-Enhanced Computed Tomography
Acronym: CINOPSIS CT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Guerbet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 1323-07-872
Record Dates: First submitted 2008-11-17; First posted 2008-11-19 (Estimated); Results first posted 2017-09-29 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-02

CONDITIONS: Renal Impairment
Keywords: Renal; Kidney; Contrast Induced Nephropathy
MeSH Terms: conditions — Renal Insufficiency | interventions — ioversol; iodixanol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Ioversol 320 mgI/mL
  Interventions: Drug: Ioversol 320 mgI/mL
- 2 (Active Comparator): Iodixanol 320 mgI/mL
  Interventions: Drug: Iodixanol 320 mgI/mL

INTERVENTIONS:
Drug: Ioversol 320 mgI/mL — 125 mL of Ioversol administered in the vein
  Other Names: Optiray
  Arms: 1
Drug: Iodixanol 320 mgI/mL — 125 mL of Iodixanol administered in the vein
  Other Names: Visipaque
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the contrast-induced nephropathy (CIN) rate in subjects randomized to receive either Ioversol or Iodixanol for contrast-enhanced computed tomography.

DETAILED DESCRIPTION:
Contrast-induced nephropathy (CIN) is an acute decline in renal function after the administration of iodinated contrast agents. CIN is commonly defined as an increase in post contrast serum creatinine (SCr) greater than or equal to 25% or an absolute increase greater than or equal to 0.5 mg/dL from pre contrast baseline values. Study will evaluate and compare the effects of two (2) contrast media products on renal function in subjects with stable reduced renal function while undergoing contrast-enhanced computed tomography.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 years of age or older
* Subjects scheduled for a clinically indicated CECT requiring 40 grams of iodine (125 mL)
* Subjects have an abnormal screening SCr that results in a calculated eGFR of < 60 mL/min/1.73 m2 using the MDRD formula and acute causes for an elevation in SCr have been excluded
* Subjects have stable reduced renal function which is defined as an abnormal screening SCr measurement with a < 15% difference from the oldest historical SCr measurement obtained within the proceeding 1 week to 12 weeks
* Subjects must provide written consent and agree to abide by the site and study requirements

Exclusion Criteria:

* Subjects previously entered into this study
* Subjects on dialysis
* Subjects received any investigational drug within 30 days of contrast administration or participated in an investigational study within 30 days prior to study enrollment
* Subjects have undergone a procedure using iodinated or gadolinium contrast agent within 7 days prior to contrast administration, or is scheduled to receive additional doses of contrast agents during the 48-72 hour post-study contrast administration
* Subjects in acute renal failure or have one or more known causes of acute renal failure
* Subjects have known or suspected unstable renal function
* Subjects scheduled for a surgical intervention or other procedure within 72 hours after the contrast administration
* Subjects taking NSAIDs (with the exception of ASA) and/or any type of diuretics who cannot discontinue these drugs post contrast administration and hold all subsequent doses until the 48-72 hour post contrast SCr has been drawn
* Subjects taking aminoglycosides
* Subjects known to have an organ transplantation
* Subjects have severe congestive heart failure (Class III-IV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eddie Darton, MD, Study Director — Mallinckrodt
Locations (13):
- United States (13):
  - UAB Hospital, Birmingham, Alabama
  - Radiology LTD, Tucson, Arizona
  - Providence Hospital, Washington D.C., District of Columbia
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Maine Research Associates, Auburn, Maine
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - University of Rochester Medical Center, Rochester, New York
  - Wake Research Associates, Raleigh, North Carolina
  - Radiology Consultants, Inc., Youngstown, Ohio
  - Geisinger Medical Center, Danville, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - Trinity Clinic, Tyler, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 6 patients signed an informed consent for the study and therefore were considered as included
Groups:
- Iodixanol: Patients randomized to receive Iodixanol 320 mgI/mL.
- Ioversol: Patients randomized to receive Ioversol 320 mgI/mL.
Period: Overall Study
Arm/Group | Iodixanol | Ioversol
Started | 2 | 4
Completed | 2 | 3
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- IodixanoI: Patients randomized to receive iodixanol 320 mgI/mL.
- IoversoI: Patients randomized to receive ioversol 320 mgI/mL.
- Total: Total of all reporting groups
Arm/Group | IodixanoI | IoversoI | Total
Number analyzed (Participants) | 2 | 4 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.8 (7.0) | 69.8 (7.0) | 69.8 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Contrast-induced Nephropathy (CIN)
Description: Contrast-induced nephropathy (CIN) is defined as an increase of ≥ 25% or an increase of ≥ 0.5 mg/dL from baseline serum creatinine (SCr), within 48 - 72 hours after contrast medium administration.
  For each patient, SCr values were measured from 2 to 24 hours before and from 48 to 72 hours after contrast medium administration.
Time Frame: Based on the SCr values of each patient measured from 2 to 24 hours before and from 48 to 72 hours after contrast medium administration
Population: One patient from the Ioversol arm was prematurely withdrawn just after contrast medium administration due to the discovery of a new brain mass. Consequently, no SCr measurement was performed for this patient and the primary outcome could not be analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- Iodixanol: Patients who received iodixanol
- IoversoI: Patients who received ioversol
Arm/Group | Iodixanol | IoversoI
Number analyzed (Participants) | 2 | 3
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: All adverse events occuring during the time from signing of informed consent to the conclusion of the study were recorded. Overall, the study duration ranged from 1 day to 86 days.
Groups:
- Iodixanol: Patients who received iodixanol 320 mgI/mL.
- Ioversol: Patients who received ioversol 320 mgI/mL.
Arm/Group | Iodixanol | Ioversol
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/2 | 1/4
Other Adverse Events (participants affected / at risk) | 1/2 | 1/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iodixanol (N=2) | Ioversol (N=4)
Asymptomatic brain mass (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Iodixanol (N=2) | Ioversol (N=4)
Diarrhea (Gastrointestinal disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Due to the small number of patients enrolled, no statistical analyses were performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No